CLINICAL TRIAL: NCT03388632
Title: Phase I Study of Recombinant Interleukin 15 in Combination With Checkpoint Inhibitors Nivolumab and Ipilimumab in Subjects With Refractory Cancers
Brief Title: Recombinant Interleukin-15 in Combination With Checkpoint Inhibitors Nivolumab and Ipilimumab in People With Refractory Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jibran Ahmed, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180033; 18-C-0033
Record Dates: First submitted 2017-12-30; First posted 2018-01-03 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Solid Tumors; Treatment-Refractory Cancers
Keywords: Immunotherapy; T Cells; Checkpoint Inhibitor; IL-15; Combination Therapy
MeSH Terms: interventions — Ipilimumab; Nivolumab; Electrocardiography; Echocardiography; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lead-in Doublet A (Experimental): Lead-in doublet for initial safety evaluation: Recombinant interleukin-15 (rhIL-15) given subcutaneous (SC) days 1-8 and 22- 29 + nivolumab (anti-programmed cell death protein 1 (PD1) given intravenous (IV) on days 8, (IL-15 doses are limited to first 4 cycles only).
  Interventions: Drug: rhIL-15; Drug: Nivolumab; Diagnostic Test: EKG; Diagnostic Test: ECHO; Diagnostic Test: CT Scan
- Lead-in Doublet B (Experimental): Lead-in doublet for initial safety evaluation: Recombinant interleukin-15 (rhIL-15) given subcutaneous (SC) days 1-8 and 22- 29 + ipilimumab (anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) given intravenous (IV) on day 8, (IL-15 doses are limited to first 4 cycles only).
  Interventions: Drug: rhIL-15; Drug: Ipilimumab; Diagnostic Test: EKG; Diagnostic Test: ECHO; Diagnostic Test: CT Scan
- Triplet C (Experimental): Dose escalation of the triplet combination: Recombinant human interleukin-15 (rhIL-15) given subcutaneous (SC) days 1-8 and 22- 29 + nivolumab (anti-programmed cell death protein 1 (PD1) given intravenous (IV) on days 8 + ipilimumab (anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) given intravenous (IV) on day 8, IL-15 will initially be given at 0.5 µg/kg/day (dose level 1, DL1). If the safety profile is acceptable at DL1, the dose of IL-15 will be increased to 1.0 µg/kg/day (DL2) in subsequent patients, then to 2.0 µg/kg/day (DL3) if the safety profile of DL2 is acceptable. (IL-15 doses are limited to first 4 cycles only).
  Interventions: Drug: rhIL-15; Drug: Ipilimumab; Drug: Nivolumab; Procedure: Tumor biopsies; Diagnostic Test: EKG; Diagnostic Test: ECHO; Diagnostic Test: CT Scan

INTERVENTIONS:
Drug: rhIL-15 — Recombinant human interleukin 15 (IL-15) is a stimulatory cytokine that activates the immune system, inducing proliferation of T lymphocytes and naturel killer (NK) cells. Administration of recombinant human IL-15 (rhIL-15) has been shown to result in a dramatic increase of circulating cytotoxic T lymphocyte (CD8+T) cells and NK cells; these changes in immune cell populations suggest potential for anti-tumor activity.
  Other Names: recombinant human interleukin 15
Drug: Ipilimumab — Ipilimumab is a fully human monoclonal antibody against cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), a receptor present on the surface of activated T cells that functions as an immune checkpoint. Immune checkpoints pathways typically act to downregulate T cell activity and are co-opted by tumors to allow the malignant cells to evade the immune response. Blocking the engagement of CTLA-4 with ipilimumab allows infiltrating T cells to mount an anti-tumor response. Ipilimumab is approved by the Food and Drug Administration (FDA) for the treatment of certain patients with melanoma and has shown clinical activity in other tumor types as well.
  Other Names: Yervoy
  Arms: Lead-in Doublet B; Triplet C
Drug: Nivolumab — Nivolumab is a humanized monoclonal antibody against programmed death 1 (PD-1), a receptor present on the surface of activated T cells that functions as an immune checkpoint. One of the ligands for PD-1, programmed death-ligand 1 (PD-L1), is commonly expressed by tumor cells. Similar to inhibition of the cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) pathway by ipilimumab, blocking of PD-1/PD-L1 signaling by nivolumab allows infiltrating T cells to mount an immune response against the tumor. Nivolumab is approved as a single agent for several cancer types, as well as for the treatment of advanced melanoma in combination with ipilimumab.
  Other Names: Opdivo
  Arms: Lead-in Doublet A; Triplet C
Procedure: Tumor biopsies — Triplet C Pre-study and Cycle 1, Week 6.
  Other Names: Tumor bx
  Arms: Triplet C
Diagnostic Test: EKG — Pre-study
  Other Names: Electrocardiogram
Diagnostic Test: ECHO — Pre-study
  Other Names: Echocardiogram
Diagnostic Test: CT Scan — Restaging every cycle (every 6 weeks) ± 1 week during cycles 1-4 and every 2 cycles (every 12 weeks) ± 1 week thereafter.
  Other Names: Computed tomography scan

SUMMARY:
Background:

The drug Interleukin-15 (IL-15) activates the immune system. The drugs nivolumab and ipilimumab unblock immune cells. The drugs together may allow immune cells to recognize and attack cancer cells, causing tumors to shrink.

Objective:

To test the effects and maximum dose of IL-15, nivolumab, and ipilimumab.

Eligibility:

People ages 18 and older who have cancer that does not respond to treatment

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Heart, blood, and urine tests
* Scans

Tumor biopsy: A small needle removes a tumor sample.

Participants will be in 1 of 3 treatment groups:

* IL-15 with nivolumab
* IL-15 with ipilimumab
* IL-15 with nivolumab and ipilimumab

Participants will take the drugs in four 6-week cycles. IL-15 is injected under the skin. The other two drugs are injected into an arm vein over 60-90 minutes. Participants may need to stay at the hospital 2-3 hours after the first dose of any drug to watch for side effects.

Each cycle will include:

* Weekly blood and urine tests
* 16 IL-15 injections
* 1 ipilimumab injection if applicable
* 3 nivolumab injections if applicable
* Blood tests weekly during cycles 1 and 2
* Urine tests weekly during cycles 1 and 2
* Scans and a tumor biopsy on day 42

After cycle 4, participants will stop taking IL-15. They will continue the other drugs until they can no longer tolerate the side effects, or their cancer gets worse. Those cycles will include:

* 1 ipilimumab injection if applicable
* 3 nivolumab injections if applicable
* Scans every other cycle

After participants stop treatment, their doctor will monitor their side effects for 4 months or until they go away.

DETAILED DESCRIPTION:
BACKGROUND:

* Interleukin-15 (IL-15) is a stimulatory cytokine that activates the immune system, inducing proliferation of T lymphocytes and natural killer (NK) cells. Administration of recombinant human IL-15 (rhIL-15) has been shown to result in a dramatic increase of circulating cytotoxic T lymphocytes (CD8+T cells) and NK cells; these changes in immune cell populations suggest potential for anti-tumor activity.
* Immune checkpoint inhibitors, including nivolumab (anti-programmed cell death protein 1 (PD-1) and ipilimumab (anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), block the engagement of specific T-cell signaling pathways by tumor cells. These regulatory pathways typically act to downregulate T cell activity and are co-opted by tumors to allow the malignant cells to evade the immune response.
* The combination of rhIL-15 with two checkpoint inhibitor therapies has potential to lead to enhanced immune activation, resulting in anti-tumor T cell responses that are effective in refractory cancers.

PRIMARY OBJECTIVE:

- Determine the safety, toxicity profile, dose-limiting toxicity (DLT) and maximum tolerated doses (MTD) of subcutaneous administration of rhIL-15 given in combination with the anti- CTLA-4 antibody ipilimumab and the anti-PD-1 antibody nivolumab in patients with metastatic or treatment-refractory cancers.

EXPLORATORY OBJECTIVE:

* Assess the clinical activity of rhIL-15, ipilimumab, and nivolumab combination therapy as characterized by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune RECIST (iRECIST) response rate of patients treated in this trial.
* Investigate the biological effects of this combination on circulating T cell subsets and on PD-1/programmed death-ligand 1 (PD-L1) expression and immune cell activation in tumor tissue.

ELIGIBILITY:

- Patients greater than or equal to 18 years of age with histologically confirmed solid tumor malignancy that is metastatic or treatment-refractory cancers.

STUDY DESIGN:

* The first 4-6 patients enrolling in the study will be placed into lead-in doublets with a combination of rhIL-15 and either nivolumab OR ipilimumab; once toxicity is cleared in both doublets (i.e., 2 patients enrolled on each doublet remain free of DLTs for 6 weeks) and a safety analysis is reviewed and approved by the Institutional Review Board (IRB), new patients will be enrolled directly onto the triple agent combination.
* For the first four 42-day cycles on the triplet, patients will receive subcutaneous (SC) rhIL-15 on days 1-8 and 22-29, intravenous (IV) nivolumab on days 8, 22, and 36, and IV ipilimumab on day 8. Cycles 5 and onwards will not include treatment with rhIL-15.
* Patients will be encouraged to report any and all adverse events, given the high likelihood of toxicities with the triplet combination therapy.
* Blood for pharmacodynamic (PD) endpoints will be collected throughout the study and tumor biopsies will be collected pretreatment and on cycle 1, day 42 (C1D42) (optional during the doublets and triplet escalation phase, mandatory during the triplet expansion phase)

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must have histologically confirmed solid tumor malignancy that is metastatic or treatment refractory cancers which are not curable or do not have known measures or treatments that are associated with a survival advantage (as defined by the subject or the physician investigator). Enrollment of subjects with tumors that can be safely biopsied is encouraged.

Subjects must have evaluable, or measurable disease defined as greater than or equal to 1 lesion that can be accurately measured in greater than or equal to 1 dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with a spiral computed tomography (CT) scan.

Subjects must have recovered to less than or equal to grade 1 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) or stabilized from toxicity of prior chemotherapy or biologic therapy administered more than 4 weeks or 5 half-lives earlier, whichever is shorter.

Subjects on bisphosphonates/denosumab for any cancer or on hormone therapy for prostate cancer may continue this therapy. However, subjects with prostate cancer must have confirmed metastatic disease that has progressed despite hormonal therapy or refused or is intolerant of hormonal therapy.

Age greater than or equal to 18 years.

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky or Lansky greater than or equal to 70%.

Subjects must have normal organ and marrow function as defined below:

* Leukocytes greater than or equal to 2,000/mm^3
* Absolute neutrophil count (ANC) greater than or equal 1,500/mm^3
* Platelets greater than or equal to 100,000/mm^3
* Total bilirubin less than or equal to 1.5 times institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to 1.5 times institutional upper limit of normal (ULN) or if liver metastasis, less than or equal to 2.5 times ULN
* Serum creatinine less than or equal to 1.5 times institutional ULN, OR Creatinine clearance greater than or equal to 50 mL/min/1.73 m^2 for subjects with serum creatinine levels greater than 1.5 times higher than institutional normal
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

Subjects with inactive central nervous system (CNS) metastasis are eligible. Inactive CNS metastasis is defined as: no symptoms of brain metastases after successful definitive treatment of brain metastases (surgical resection, whole brain irradiation, stereotactic radiation therapy, or a combination of these) with stable or improved radiographic appearance on magnetic resonance imaging (MRI) scan at least 1 month after completion of treatment.

Subjects may have previously progressed on treatment with one of the 3 agents being used in this trial or treatment with other checkpoint inhibitors, as long as they have recovered from previous toxicity. Subjects that previously progressed on treatment with a combination of any 2 of the 3 agents being used in this trial are eligible for the triplet cohort only.

The effects of ipilimumab, nivolumab, and rhIL-15 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the treatment portion of the study, and for a minimum for 5 months (women) and 7 months (men) after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Ability to understand and the willingness to sign a written informed consent document.

Willingness to provide blood and biopsy samples for research purposes if on the expansion phase of the study.

EXCLUSION CRITERIA:

Subjects who have received any prior cytotoxic therapy, immunotherapy, major surgery, antitumor vaccines or monoclonal antibodies in the 4 weeks or 5 half-lives, whichever is shorter, prior to cycle 1, day 1 (C1D1) (6 weeks prior for checkpoint inhibitors such as anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) or anti-programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PD-L1) and for nitrosoureas or mitomycin C). Subjects must not have received radiotherapy in the 2 weeks prior to C1D1. Subjects who had grade greater than or equal to 3 immune-related adverse events (irAE) (excluding endocrinopathies) during previous treatment with one of the checkpoint inhibitors are excluded from the trial; subjects who had grade 1 or 2 irAE (including serious AEs) that have resolved to grade 1 are eligible at the discretion of the principal investigator (PI).

Subjects with primary brain cancers or active central nervous system (CNS) metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the agents on this trial.

Concurrent anticancer therapy (including other investigational agents) with the exception of hormone therapy for breast or prostate cancer. Patients that have received treatment for a different cancer previously and have been disease-free for less than one year are excluded.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cognitive impairment, active substance abuse, or psychiatric illness/social situations that, in the view of the Investigator, would preclude safe treatment or the ability to give informed consent and limit compliance with study requirements.

Inability or refusal to practice effective contraception during therapy or the presence of pregnancy or active breastfeeding. Because there is no significant preclinical information regarding the risk to a fetus or newborn infant, pregnant or breastfeeding women will be excluded from participation in this trial.

Documented human immunodeficiency virus (HIV) infection or positive serology. Since rhIL-15 treatment stimulates the subject's immune system to attack their tumor, the defective immune systems of subjects with HIV makes responses to this treatment much less likely to provide benefit and these subjects are not eligible for this trial.

History of severe asthma (subjects with a history of mild asthma that are on or can be switched to non-corticosteroid bronchodilator regimens are eligible).

Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. The use of inhaled corticosteroids is allowed.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jibran Ahmed, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data in a National Institutes of Health (NIH) - funded or approved public repository, identified data in the Biomedical Translational Research Information System (BTRIS) (automatic for activities in the NIH Clinical Center), and de-identified or identified data with approved outside collaborators under appropriate agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the time of publication or shortly thereafter.
Access Criteria: Data will be shared through a National Institutes of Health (NIH) - funded or approved public repository: clinicaltrials.gov, Biomedical Translational Research Information System (BTRIS) (automatic for activities in the NIH Clinical Center), approved outside collaborators under appropriate individual agreements, and publication and/or public presentations.

REFERENCES:
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Lipson EJ, Drake CG. Ipilimumab: an anti-CTLA-4 antibody for metastatic melanoma. Clin Cancer Res. 2011 Nov 15;17(22):6958-62. doi: 10.1158/1078-0432.CCR-11-1595. Epub 2011 Sep 7. PMID 21900389
- [Background] Conlon KC, Lugli E, Welles HC, Rosenberg SA, Fojo AT, Morris JC, Fleisher TA, Dubois SP, Perera LP, Stewart DM, Goldman CK, Bryant BR, Decker JM, Chen J, Worthy TA, Figg WD Sr, Peer CJ, Sneller MC, Lane HC, Yovandich JL, Creekmore SP, Roederer M, Waldmann TA. Redistribution, hyperproliferation, activation of natural killer cells and CD8 T cells, and cytokine production during first-in-human clinical trial of recombinant human interleukin-15 in patients with cancer. J Clin Oncol. 2015 Jan 1;33(1):74-82. doi: 10.1200/JCO.2014.57.3329. Epub 2014 Nov 17. PMID 25403209
- [Derived] Waldmann TA, Dubois S, Miljkovic MD, Conlon KC. IL-15 in the Combination Immunotherapy of Cancer. Front Immunol. 2020 May 19;11:868. doi: 10.3389/fimmu.2020.00868. eCollection 2020. PMID 32508818
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0033.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg: Doublet A, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29 and Nivolumab intravenous (IV) d8, 22, & 36. DOUBLET A: Cycle 1-4, IL-15: 0.5 mcg/kg subcutaneously d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36; Cycle 5+ Nivolumab 240 mg IV over 60 min d1, 15 & 29.
- Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg: Doublet A, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29 and Nivolumab intravenous (IV) d8, 22, & 36. Cycles 5+, Nivolumab alone (IV d1, 15 & 29) after Doublet A. DOUBLET A: Cycle 1-4, IL-15: 0.5 mcg/kg subcutaneously d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36; Cycle 5+ Nivolumab 240 mg IV over 60 min d1, 15 & 29.
- Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg: Doublet B, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29 and Ipilimumab intravenous (IV) d8. DOUBLET B: Cycle 1-4, IL-15: 0.5 mcg/kg subcutaneously on d1-8 & 22-29 plus Ipilimumab 1 mg/kg IV over 90-minute (min) d8; Cycle 5+ Ipilimumab 1 mg/kg IV over 90 min d1.
- Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg: Triplet, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29, Nivolumab intravenous (IV) d8, 22, & 36 and Ipilimumab IV d8. TRIPLET 1: Cycle 1-4, IL-15: 0.5 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1.
- Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg: Triplet, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29, Nivolumab intravenous (IV) d8, 22, & 36 and Ipilimumab IV d8. TRIPLET 2: Cycle 1-4, IL-15: 1 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1.
- Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg: Triplet, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29, Nivolumab intravenous (IV) d8, 22, & 36 and Ipilimumab IV d8. TRIPLET 3: Cycle 1-4, IL-15: 2 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1.
- Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg: Triplet, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29, Nivolumab intravenous (IV) d8, 22, & 36 and Ipilimumab IV d8. TRIPLET 3: Cycle 1-4, IL-15: 2 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1. TRIPLET 2: Cycle 1-4, IL-15: 1 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1.
- Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg: Triplet, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29, Nivolumab intravenous (IV) d8, 22, & 36 and Ipilimumab IV d8. Triplet, cycles 5+ Nivolumab IV d1, 15, & 29 and Ipilimumab IV d1. TRIPLET 1: Cycle 1-4, IL-15: 0.5 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1.
- Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg: Triplet, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29, Nivolumab intravenous (IV) d8, 22, & 36 and Ipilimumab IV d8. Triplet, cycles 5+ Nivolumab IV d1, 15, & 29 and Ipilimumab IV d1. TRIPLET 2: Cycle 1-4, IL-15: 1 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1.
Period: Lead-In Doublet A
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg
Started | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Lead-In Doublet B
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg
Started | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Triplet C
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg
Started | 0 | 0 | 0 | 2 | 18 | 2 | 1 | 2 | 1
Completed | 0 | 0 | 0 | 2 | 16 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — 42-day lapse in tx | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Switched to alternative treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant choice | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Total
Number analyzed (Participants) | 2 | 1 | 2 | 2 | 18 | 2 | 1 | 2 | 1 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 2 | 15 | 2 | 1 | 2 | 1 | 27
  >=65 years | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.02) | 49 (0) | 51 (26.87) | 53 (1.41) | 56.14 (12.04) | 52 (11.31) | 55 (0) | 49 (4.24) | 60 (0) | 54.55 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 12 | 0 | 1 | 2 | 1 | 18
  Male | 2 | 1 | 1 | 1 | 6 | 2 | 0 | 0 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 2 | 1 | 2 | 2 | 15 | 2 | 1 | 2 | 1 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 6
  White | 1 | 1 | 1 | 1 | 13 | 1 | 0 | 2 | 1 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 2 | 2 | 18 | 2 | 1 | 2 | 1 | 31

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) at Which Dose-Limiting Toxicities (DLT) Occurred With rhIL-15 Administered in Combination With Fixed Doses of Nivolumab and Ipilimumab
Description: Here is the maximum tolerated dose (MTD) (i.e., highest dose) of rhIL-15 administered in combination with fixed doses of nivolumab and ipilimumab at which dose-limiting toxicities occurred in ≤1 of 6 participants during cycle 1, dose escalation in participants receiving the triplet combination. A DLT is defined as an adverse event that is felt to be related (possibly, probably, or definitely) to administration of study drugs, and meets prespecified criteria, including any condition requiring long-term treatment with corticosteroids or permanent discontinuation of one of the agents.
Time Frame: Cycle 1 (42 days)
Population: This analysis includes participants (pts) from multiple groups, as different groups received different doses of rhIL-15. Includes pts from group 4 (n=2), group 5 (n=9), group 6 (n=2), group 7 (n=1), group 8 (n=2), and group 9(n=1). Of the 18 pts in group 5, 9 pts were enrolled in the dose escalation phase to determine MTD & an additional 9 pts were enrolled in an expansion cohort at that dose after the MTD was determined. Pts in this expansion cohort were not included in the MTD determination.
Measure: Number; unit: mcg/kg/day
Groups:
- All Participants in Escalation Phase of Arm C: All participants who received at least one dose of rh IL-15 subcutaneously administered in combination with fixed doses of nivolumab and ipilimumab on cycle 1 (42 days).
Arm/Group | All Participants in Escalation Phase of Arm C
Number analyzed (Participants) | 17
mcg/kg/day | 1.0

2. Primary Outcome: Number of Dose-limiting Toxicities (DLT) Possibly, Probably, or Definitely Related to Study Drugs
Description: A DLT is defined as an adverse event (AE) that is felt to be related (possibly, probably, or definitely) to administration of study drugs, and meets prespecified criteria, including any condition requiring long-term treatment with corticosteroids or permanent discontinuation of one of the agents.
Time Frame: Cycle 1 (42 days)
Population: As pre-specified in the protocol, DLT's were assessed in the lead-in doublet arms and the triplet escalation phase groups only.
Measure: Number; unit: toxicities
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg
Number analyzed (Participants) | 2 | 1 | 2 | 2 | 18 | 2 | 1 | 2 | 1
toxicities
  Possibly related to rh IL-15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Probably related to rh IL-15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Definitely related to rh IL-15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Possibly related to Nivolumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Probably related to Nivolumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Definitely related to Nivolumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Possibly related to Ipilimumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Probably related to Ipilimumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Definitely related to Ipilimumab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLT)
Description: Here is the number of participants experiencing dose-limiting toxicities (DLT). A DLT is defined as an adverse event that is felt to be related (possibly, probably, or definitely) to administration of study drugs, and meets prespecified criteria, including any condition requiring long-term treatment with corticosteroids or permanent discontinuation of one of the agents.
Time Frame: Cycle 1 (42 days)
Population: Of the 18 participants in group 5, 9 participants were enrolled in the dose escalation phase to determine maximum tolerated dose (MTD), and an additional 9 participants were enrolled in an expansion cohort at that dose after the MTD was determined. Participants in this expansion cohort were not included in this DLT evaluation per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg: Triplet, cycles 1-4: Recombinant Human Interleukin (rH IL-15) subcutaneous (SC) day(d)1-8 & 22-29, Nivolumab intravenous (IV) d8, 22, & 36 and Ipilimumab IV d8. TRIPLET 3: Cycle 1-4, IL-15: 2 mcg/kg subcutaneously on d1-8 & d22-29 plus Nivolumab 240 mg IV over 60-minute (min) d8, 22, & 36 and Ipilimumab 1 mg/kg IV over 90 min d8; Cycle 5+ Nivolumab 240 mg IV over 60 min on d1, 15 & 29 plus Ipilimumab 1 mg/kg IV over 90 min d1.
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg
Number analyzed (Participants) | 2 | 1 | 2 | 2 | 9 | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events were monitored/assessed from the first study intervention through 30 days after the study agent (s) was/were administered up to approximately 23 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg
Number analyzed (Participants) | 2 | 1 | 2 | 2 | 18 | 2 | 1 | 2 | 1
Participants | 2 | 1 | 2 | 2 | 18 | 2 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed up to approximately 23 months. Adverse Events were monitored/assessed from the first study intervention through 30 days after the study agent (s) was/were administered up to approximately 23 months.
Arm/Group | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/2 | 0/2 | 1/18 | 0/2 | 0/1 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 0/1 | 1/2 | 2/2 | 13/18 | 2/2 | 1/1 | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 2/2 | 2/2 | 18/18 | 2/2 | 1/1 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg (N=2) | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg (N=1) | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg (N=2) | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=2) | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=18) | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg (N=2) | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=1) | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=2) | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg (N=1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complicated kidneystone removal procedure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion-related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg (N=2) | Arm A/Arm A1 Doublet A - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Nivolumab 240mg (N=1) | Arm B Doublet B - Recombinant Human Interleukin (rH IL-15) 0.5mcg/kg & Ipilimumab 1mg/kg (N=2) | Arm C Triplet 1-Recombinant Human Interleukin(rHIL-15) 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=2) | Arm C Triplet 2-Recombinant Human Interleukin(rHIL-15) 1mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=18) | Arm C Triplet 3-Recombinant Human Interleukin(rHIL-15) 2mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg (N=2) | Arm C Triplet 3/Triplet 2/Recombinant Human Interleukin 2mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=1) | Arm C/Arm C1 Triplet 1 - Recombinant Human Interleukin 0.5mcg/kg/Nivolumab 240mg/Ipilimumab 1mg/kg (N=2) | Arm C/Arm C1 Triplet 2-Recombinant Human Interleukin 1mcg/kg & Nivolumab 240mg/Ipilimumab 1mg/kg (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (3) | 1 (4) | 0 (0) | 7 (15) | 1 (1) | 1 (5) | 1 (7) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 2 (4) | 1 (1) | 7 (12) | 1 (2) | 0 (0) | 2 (6) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (6) | 1 (1) | 15 (57) | 0 (0) | 0 (0) | 1 (33) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 9 (14) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 1 (4) | 0 (0) | 10 (23) | 1 (1) | 1 (4) | 1 (11) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 5 (9) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (11) | 0 (0) | 1 (12) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 14 (23) | 2 (2) | 1 (1) | 2 (7) | 1 (4)
Cholesterol high (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 1 (15) | 1 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (2) | 1 (1) | 4 (6) | 1 (2) | 1 (2) | 1 (4) | 1 (4)
CPK increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (4) | 1 (3) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (3) | 1 (1) | 1 (3)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (8) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 4 (4) | 1 (2) | 0 (0) | 1 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Edema limbs (General disorders) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify: Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify: TSH increase (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify: Kaleidescopic vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Eye disorders - Other, specify: black eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify: stye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 11 (18) | 0 (0) | 1 (1) | 2 (13) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0) | 1 (2) | 2 (4) | 12 (27) | 2 (2) | 1 (2) | 2 (2) | 1 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify: belching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (2) | 1 (4) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 4 (5) | 0 (0) | 1 (2) | 2 (10) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (8) | 1 (1) | 2 (3) | 2 (2) | 13 (21) | 2 (2) | 1 (5) | 2 (12) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (5) | 1 (4) | 1 (10) | 1 (1) | 11 (23) | 1 (1) | 1 (1) | 2 (29) | 1 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (5) | 1 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (2) | 2 (5) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 7 (12) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 3 (8) | 0 (0) | 1 (2) | 1 (8) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (9) | 12 (22) | 1 (2) | 0 (0) | 2 (13) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify: thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 1 (7) | 1 (3) | 2 (4) | 13 (20) | 2 (2) | 1 (4) | 2 (7) | 1 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactate dehydrogenase increased (Investigations) | 1 (3) | 1 (1) | 2 (2) | 0 (0) | 7 (12) | 1 (1) | 1 (3) | 0 (0) | 1 (7)
Lipase increased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 5 (19) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 1 (7) | 0 (0) | 1 (1) | 8 (18) | 0 (0) | 0 (0) | 1 (1) | 1 (8)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: Upper back spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: cramp in legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify: tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (7) | 1 (1) | 1 (5) | 1 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 2 (4) | 5 (13) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (9) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (25) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (4) | 0 (0) | 1 (4) | 0 (0) | 10 (19) | 1 (1) | 0 (0) | 1 (10) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 1 (6) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify: Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify: protein/creatine ratio increase (Renal and urinary disorders) | 1 (4) | 0 (0) | 2 (5) | 1 (2) | 6 (10) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify: Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Serum amylase increased (Investigations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (5) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 8 (13) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Rash Dermatitis NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Dermatitis NOS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Lipoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — : Rash dermatitis serum sickness-like reaction
Skin and subcutaneous tissue disorders - Other, specify: abrasion scrotum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: chest rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify: erythematous macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify: compli kidney stone removal prod (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (11) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Weight loss (Investigations) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (2) | 1 (5) | 2 (3) | 7 (23) | 0 (0) | 0 (0) | 1 (21) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT03388632/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Triplet Consent (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03388632/ICF_001.pdf
  • Informed Consent Form: Standard Doublet Consent (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT03388632/ICF_002.pdf